CLINICAL TRIAL: NCT03963024
Title: Treosulfan and Total-marrow Irradiation (TMI) Based Conditioning With Rapamycin Based Graft vs. Host Disease (GvHD) Prophylaxis for Allogenic Stem Cell Transplantation (Allo-HSCT) in Patients With High-risk Hematological Malignancies
Brief Title: Treosulfan-TMI Conditioning and Rapamycin GvHD Prophylaxis Before Allo-HSCT
Acronym: TrRaMM-TMI
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: low rate of enrolment
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Ciceri Fabio, Professor, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-002479-16
Record Dates: First submitted 2019-05-21; First posted 2019-05-24 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Irradiated Bone Marrow; Transplant-Related Hematologic Malignancy; Leukemia, Acute; Multiple Myeloma; Graft Vs Host Disease
MeSH Terms: conditions — Leukemia; Multiple Myeloma; Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm Treatment (Experimental): Conditioning treatment "Treosulfan+TMI"; SCT; GvHD prophylaxis;
  Interventions: Drug: Conditioning treatment "Treosulfan-TMI"; Procedure: SCT; Drug: GvHD prophylaxis

INTERVENTIONS:
Drug: Conditioning treatment "Treosulfan-TMI" — Treosulfan i.v.: 14 g/m²/d (day -6 to -4) Fludarabine i.v.: 30 mg/m²/d (day -6 to -2) Antithymocyte globulin (ATG)-Fresenius i.v.: 5/0 mg/kg (day -4 to -2) Mabthera i.v.: 200/0* mg/m2 (day -1) TMI: (10 Gy) 2 Gy bis in die (BID) (day -2 to -1) or TMI: (12 Gy) 2 Gy BID (day -3 to -1) or TMI: (14 Gy) 2 Gy BID (day -3 to -1)
Procedure: SCT — Stem Cell Transplant
Drug: GvHD prophylaxis — Rapamycin p.o.: 4 mg/d, (target 8-15 ng/ml) (starting day -7) Mycofenolate mofetile: 10 mg/kg tid, (Maximum dose 720 mg/tid) (starting from day 0)

SUMMARY:
TrRaMM-TMI is a phase I trial to evaluate the feasibility and efficacy of an original sequential TMI/TrRaMM (Total Marrow Irradiation/Treosulfan-Rapamycin-Mycophenolate Mofetil) schedule in patients with hematological malignancies in advanced stage of disease undergoing an allogenic Stem Cell Transplant (SCT).

The aim is to determine the maximum tolerated dose of TMI when combined with conditioning chemotherapy to transplant according to TrRaMM schedule.

ELIGIBILITY:
Inclusion Criteria:

* Patients with haematological malignancies such as

  * any acute myeloid leukemia (AML) beyond Complete Remission (CR) 1
  * any acute lymphoblastic leukemia (ALL) beyond CR1
  * multiple myeloma (MM) at any relapse/progression, except refractory disease
  * MM with unfavourable cytogenetic profile at diagnosis
  * MM with less than a partial response (PR) after induction therapy
* Karnofsky Index ≥ 80 %
* Adequate contraception in female patients of child-bearing potential.
* Written informed consent
* Availability of one of the following:

  * A matched related or unrelated donor (MRD or MUD)

Exclusion Criteria:

* A hematopoietic cell transplantation-specific comorbidity index > 4
* Active non-controlled infectious disease at the moment of inclusion
* Active hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Impaired liver function (Bilirubin > 2.0 x upper normal limit; Transaminases > 3.0 x upper normal limit)
* Impaired renal function (Creatinine-clearance < 60 ml/min; Serum Creatinine > 1.5 x upper normal limit).
* Pleural effusion or ascites > 1.0 L
* Pregnancy or lactation
* Known hypersensitivity to treosulfan and/or fludarabine and/or rapamycin
* Non-co-operative behaviour or non-compliance
* Psychiatric diseases or conditions that might impair the ability to give informed consent
* Previous spinal cord radiotherapy with dose ≥ 45 Gy equivalent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2014-02-12 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of the maximum tolerated dose of TMI (FEASIBILITY of TMI) | From administration of TMI (-5) to transplant
  To determine the maximum tolerated dose of TMI when combined with conditioning chemotherapy to transplant according to TrRaMM schedule
Rate of Survival post transplant | +30 days post transplantation
  Evaluation of survival and engraftment

SECONDARY OUTCOMES:
Efficacy - progression free survival (PFS) | End of total follow-up is 365 days after transplantation of the last patient included
  PFS
Efficacy - Overall survival (OS) | End of total follow-up is 365 days after transplantation of the last patient included
  OS
Efficacy - Relapse incidence (RI) | End of total follow-up is 365 days after transplantation of the last patient included
  RI
Evaluation of Transplant Safety - incidence of non-relapse mortality (NRM) | Eon day +28, day +100 and +360
  Evaluation of incidence of NRM
Evaluation of Transplant Safety | End of total follow-up is 365 days after transplantation of the last patient included
  Cumulative of incidence and cumulative severity of GvHD

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Raffaele, Milan, Lombardy, Italy